CLINICAL TRIAL: NCT01285869
Title: Impact of a Multidimensional Intervention in Elderly Patients With Pneumonia: a Prospective Randomized Controlled Trial.
Brief Title: Impact of a Multidimensional Intervention in Elderly Patients With Pneumonia
Acronym: IMIEPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIBSP-INT-2010-13
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Community-acquired Pneumonia; Healthcare-associated Pneumonia
Keywords: Pneumonia; Intervention Studies; Aged; Aged, 80 and over; Geriatric Assessment
MeSH Terms: conditions — Community-Acquired Pneumonia; Healthcare-Associated Pneumonia; Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multidisciplinar intervention (Experimental): Patients that will receive the multidimensional intervention during the ambulatory follow-up.
  Interventions: Other: Multidimensional intervention
- Conventional follow up (No Intervention): This is an observation only group and outpatient follow up will be indicated in accordance with usual and customary practices.

INTERVENTIONS:
Other: Multidimensional intervention — The patient will be cited 2 months after hospital discharge for a geriatric evaluation carried out by a geriatric nurse and an internist with geriatric training. The duration of the first visit is 45-60 minutes. The visit consists of: 1. Assessment of the pneumonia resolution, co-morbidities, aspiration risk, risk of multiresistant infections, and the immunization, functional and cognitive status. 2. An individualized intervention plan. The patient and family or caregiver will receive an educational intervention, a written report with the planned intervention and an educational leaflet. Those patients who require further assessment or follow up of the intervention will receive 1 or 2 more visits and all the patients will be cited one year after the first visit.
  Other Names: Comprehensive geriatric assesment
  Arms: Multidisciplinar intervention

SUMMARY:
The hypothesis of this study is that long-term outcome in elderly patients admitted with the diagnosis of community-acquired pneumonia (CAP) or healthcare-associated pneumonia (HCAP) would improve with a multidimensional intervention including assessment of co-morbidities, nutritional, functional and cognitive status and immunization.

DETAILED DESCRIPTION:
Detailed description published in "Revista Española de Geriatría y Gerontología" (see citation and link)

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (aged 65 years and over), of either sex, not dependent for basic activities of daily living (Barthel index ≥60 points).
* Diagnosed with community-acquired pneumonia at the Emergency Department or Day Hospitals at "Hospital de la Santa Creu I Santa Pau"
* Admitted to hospital.

Exclusion Criteria:

* Derived from other acute care hospitals.
* Patients with HIV infection.
* Neutrophil counter<1000/mm3
* Transplanted patients.
* Barthel index<60 points.
* Terminal disease.
* No signed informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 314 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Healthcare resources utilization (readmissions and consultations to hospital and emergency department). | 1 year after hospital admission for pneumonia
  To achieve the variables related to the healthcare resource utilization, computarized medical records will be reviewed and all patients will be followed up by telephone interview one year after discharge.The cause for readmission will be recorded.

SECONDARY OUTCOMES:
Functional status | 1 year after hospital admission for pneumonia
  Data will be obtained by review of medical records and telephone interview one year after discharge.
  Dependency in basic activities of daily living will be scored using the Barthel Index (Mahoney & Barthel. Maryland State Med J 14; 61-65) which measures the capacity to perform ten basic activities and gives a quantitative estimation of the patient level of dependency, scoring to 0 (totally dependent) to 100 (totally independent).
Institutionalization | 1 year after hospital admission for pneumonia
  Data will be obtained by review of medical records and telephone interview one year after discharge.
Survival | 1 year after hospital admission for pneumonia
  Data will be obtained by review of medical records and telephone interview to patient or relatives one year after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Olga H Torres, Phd, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Domingo Ruiz, MD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Background] Torres OH, Gil E, Comas MT, Saez ME, Clotet S, Ramirez HD, Mateo M, Ruiz D. [Impact of a multidimensional intervention in elderly patients with community-acquired pneumonia: IMIEPCAP clinical trial]. Rev Esp Geriatr Gerontol. 2016 Jan-Feb;51(1):37-43. doi: 10.1016/j.regg.2015.09.004. Epub 2015 Oct 30. Spanish. PMID 26526565
- See also: Link to the article with description of the study is provided — http://www.elsevier.es/es-revista-revista-espanola-geriatria-gerontologia-124-linkresolver-impacto-una-intervencion-multidimensional-pacientes-S0211139X15001808